



## Kaiser Permanente Northern California

Institutional Review Board FWA# 00002344 IRB# 00001045

1800 Harrison Street, 10th Floor Oakland, CA 94612 (510) 625-4588 KPNC.IRB@kp.org

**DATE:** September 7, 2022

TO: Lisa Gilliam, MD, PhD

**FROM:** Kaiser Permanente Northern California IRB

**PROJECT TITLE:** [1857661-2] Overcoming therapeutic inertia among adults recently

diagnosed with Type 2 Diabetes

**REFERENCE #:** 

**SUBMISSION TYPE:** Amendment/Modification

**ACTION:** RESEARCH - NOT HSR

**DECISION DATE:** September 7, 2022 **REVIEW TYPE:** Administrative Review

**ADMINISTRATIVE CHECK-** Not applicable

IN DUE DATE:

Dear Dr. Lisa Gilliam:

On September 7, 2022, the Kaiser Permanente Northern California (KPNC) Institutional Review Board determined that your project is Not Human Subjects Research as defined by federal regulations and institutional policies (45CFR46.102).

The activity does not meet the regulatory definition of research at 45 CFR 46.102(d):

Research means a systematic investigation, including research development, testing and evaluation, designed to develop or contribute to generalizable knowledge.

Note: The word "research" should not appear in any posters or publications resulting from this project. Also, the word "clinical trial" should not appear in any posters or publications resulting from this project. Lastly, the study team may not store any identifiable data or conduct any future research use without IRB review and approval.

This determination is based on the information provided to the IRB. If the scope or nature of the project changes in a manner that could impact this review, you are required to notify the IRB Office prior to implementing this change.

You are expected, however, to implement your study or project in a manner congruent with accepted professional standards and ethical guidelines as described in the Belmont Report

(http://www.hhs.gov/ohrp/humansubjects/guidance/belmont.html).

Additionally, you are responsible for keeping a copy of this determination letter in your project files as it may be necessary to demonstrate that your project was properly reviewed.

Provide this approval letter to the Physician in Charge (PIC), Area Manager, and/or Chief of Service, to determine whether additional approvals are needed.

If you have any questions, please contact the KPNC IRB at <a href="KPNC.IRB@kp.org">KPNC.IRB@kp.org</a>. Please include your project title and reference number in all correspondence with this committee.

Sincerely,

Kaiser Permanente Northern California IRB